CLINICAL TRIAL: NCT05896722
Title: Evaluation of Core Muscle Endurance, Upper Extremity Muscle Strength, Grip Strength, and Hand-eye Coordination in Young Adults With Generalized Joint Hypermobility
Brief Title: "Core" Muscle Endurance, Upper Extremity Muscle Strength, Grip Strength, and Hand-eye Coordination in Generalized Joint Hypermobility
Status: Completed | Type: Observational
Sponsor: Bezmialem Vakif University (Other)
Responsible Party: Principal Investigator, Deniz Tuncer, Assistant professor, Bezmialem Vakif University
Other Study IDs: DT-03
Record Dates: First submitted 2023-05-08; First posted 2023-06-09 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Hypermobility, Joint; Muscle Weakness; Coordination Lack
MeSH Terms: conditions — Joint Instability; Muscle Weakness; Ataxia | interventions — Hand Strength; Pinch Strength

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: 27 young adults aged 17-26 who scored 4 or more according to the Beighton scoring
  Interventions: Other: Core muscle endurance; Other: Upper extremity muscle strength; Other: Grip strength; Other: Pinch strength; Other: Alternate hand-wall toss test
- Control group: 27 young adults aged 17-26 who scored less than 4 points according to the Beighton scoring
  Interventions: Other: Core muscle endurance; Other: Upper extremity muscle strength; Other: Grip strength; Other: Pinch strength; Other: Alternate hand-wall toss test

INTERVENTIONS:
Other: Core muscle endurance — Trunk flexion, trunk extension, side bridge exercises and prone bridge test developed by McGill will be used to evaluate core muscle endurance.
Other: Upper extremity muscle strength — Isometric muscle strength assessment of the shoulder, elbow and wrist muscles will be performed with a hand-held dynamometer.
Other: Grip strength — Grip strength will be evaluated with a hand dynamometer in the position recommended by the American Association of Hand Therapists.
Other: Pinch strength — Pinch strength will be evaluated with a pinchmeter in three positions.
Other: Alternate hand-wall toss test — To measure hand-eye coordination, it is performed by changing hands by throwing and catching the ball against the wall.

SUMMARY:
Every individual with joint hypermobility may not apply to a health institution because they do not have a complaint that will affect their daily life. Although hypermobility is a common clinical entity in the society, this issue has not been fully understood yet. In particular, individuals with GJH are either neglected in physiotherapy and rehabilitation evaluations and practices, or they encounter an incomplete assessment and physiotherapy practices. In this study, in order to better understand the effect of GJH on "core" muscle endurance, upper extremity strength, grip strength and coordination, we will include the individuals identified GJH among the university students (hypermobility severity ≥4/9 according to Beighton diagnostic criteria) as study group and the healthy peers as control group. We believe the results we will obtain at the end of our study will make a contribution to the literature in terms of revealing the role of "core" muscle endurance and upper extremity strength, grip strength and coordination in the evaluation and rehabilitation of individuals with GJH. In addition, it will contribute to the inclusion of individuals with GJH who are professional athletes, dancers or musicians in a more comprehensive evaluation program and the creation of physiotherapy and rehabilitation programs.

According to the information we have obtained from the literature, it is a fact that hypermobility can increase the susceptibility to musculoskeletal system diseases. For this reason, early solutions to problems can be provided by evaluating hypermobility in patients who apply to health institutions with various musculoskeletal complaints, raising awareness of patients with hypermobility to prevent injuries caused by hypermobility, and strengthening muscles.

DETAILED DESCRIPTION:
Many people may have more than one hypermobile joint, and when certain conditions are met, this condition called generalized joint hypermobility (GJH) is not detrimental. In recent years, the spectrum of the disorder has been changed in the classification of joint hypermobility, from asymptomatic GJH to the multisystem involvement and painful condition called hypermobile Ehlers Danlos Syndrome. Beighton criteria are most commonly used in the diagnosis of hypermobility. The Beighton score is an easy scoring method that is scored by performing five maneuvers and includes a total of nine points. If four of these maneuvers are positive, the patient is considered to have hypermobility. Numerous studies associate hypermobility with conditions such as soft tissue injuries, pain, joint instability, decreased soft tissue strength, increased frequency of traumatic injuries, and pain-related inactivity.

The study was designed as a cross-sectional descriptive and comparative study. With this study, in order to better understand the effect of GJH on core muscle endurance, upper extremity strength, grip strength, and coordination, we aim to include volunteers with identified GEH among the university students (hypermobility severity ≥4/9 according to Beighton diagnostic criteria). 27 students between the ages of 17-26 who are studying at the Faculty of Health Sciences of Bezmialem Vakif University and scored 4 and above according to the Beighton score, and the 27 students who are in the same age group studying at the same faculty, do not have GJH will be included. In the study, after evaluating flexibility with sit-reach test, core muscle endurance, upper extremity muscle strength, hand grip strength, finger grip strength and hand-eye coordination tests will be applied to all participants. SPSS v.20 program will be used for data analysis. All data will be analyzed with the Kolmogorov-Smirnov test to determine the distribution characteristics. In the study, descriptive statistics (mean±standard deviation, minimum-maximum, number and percentile) will be given for discrete and continuous variables. When the differences between two independent groups are evaluated, "t-Test in Independent Groups" in case the parametric test prerequisites are met; If not, the "Mann Whitney -U Test" will be used. "Chi-Square Test" will be used to determine the relationships between two discrete variables. When the variables meet the parametric test prerequisites, the correlation coefficients and statistical significance will be calculated with the "Pearson Test", when they do not, the correlation coefficients and statistical significance for the relations between the variables will be calculated with the "Spearman Test".

Although there are studies in the literature evaluating muscle strength, grip strength and trunk endurance in individuals with joint hypermobility, no study evaluating hand-eye coordination has been encountered. However, no study has been encountered that evaluated core muscle endurance, upper extremity strength, grip strength, and hand-eye coordination in individuals with GJH. We believe that the results we will obtain at the end of our study will contribute to the literature in terms of revealing the role of core muscle endurance and upper extremity strength, grip and coordination in the evaluation and rehabilitation of individuals with GJH.

ELIGIBILITY:
Inclusion Criteria:

* Getting a score of 4 or higher according to the Beighton criteria
* Being between the ages of 17-26

Exclusion Criteria:

* Presence of benign joint hypermobility syndrome
* Presence of any neurological, rheumatic, musculoskeletal, metabolic and connective tissue disease
* History of fracture in the upper extremity
* History of pain, deformity or surgery associated with the vertebral column and upper extremity
* Presence of cognitive, mental and/or serious psychiatric illness
* Participating in any exercise program or sportive activity in the last six months

Ages: 17 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Young adults between the ages of 17-26 years with a score of 4 or higher according to the Beighton criteria.
Sampling Method: Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-18 (Actual)

PRIMARY OUTCOMES:
Alternate hand-wall toss test | One day
  To measure hand-eye coordination, it is performed by changing hands by throwing and catching the ball against the wall. The action is repeated for a period of 30 seconds.
Core muscle endurance tests | One day
  Trunk flexion, trunk extension, side bridge exercises and prone bridge test developed by McGill will be used to evaluate core muscle endurance.

SECONDARY OUTCOMES:
Upper extremity muscle strength measurement | One day
  Isometric muscle strength assessment of the shoulder, elbow and wrist muscles will be performed with a hand-held dynamometer.
Grip strength measurement | One day
  Grip strength will be evaluated with a hand grip dynamometer in the position recommended by the American Association of Hand Therapists.
Pinch strength measurement | One day
  It will be evaluated with a pinchmeter. Measurements will be made bilaterally in three different positions as lateral, palmar and fingertip grips.

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Tuncer, PhD, PT, Principal Investigator — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)